CLINICAL TRIAL: NCT01560364
Title: Bundle Evaluation in Extra Renal Epuration, Incidence of Thrombosis
Acronym: BEERT
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0106
Record Dates: First submitted 2011-10-17; First posted 2012-03-22 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Adults Receiving Renal Replacement Therapy
Keywords: Renal replacement therapy; Hemofilter clotting; Clotting risk factor; Hemofilter clotting prevention
MeSH Terms: interventions — Renal Replacement Therapy

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hemofilter
  Interventions: Other: renal replacement therapy

INTERVENTIONS:
Other: renal replacement therapy — Prospective observational clinical multicentric study in ICU with acute renal failure requiring renal replacement therapy.

SUMMARY:
This is a prospective observational clinical multicentric study in ICU with acute renal failure requiring renal replacement therapy.

DETAILED DESCRIPTION:
Prospective before / after observational clinical multicentric study on ICU acute kidney injury during renal replacement therapy. Evaluation of incidence and exposure to hemofilter clotting.

The after phase will consist in medical measures (help for prescription) and paramedical measures (stop the filtration flow during the patient's mobilization).

ELIGIBILITY:
Inclusion Criteria:

* Adult (age > 18 years)
* Renal replacement therapy (continuous veino-veinous hemofiltration or continuous veino-veinous hemodiafiltration)
* Consent of patients

Exclusion Criteria:

* Use citrate anticoagulation
* Age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults receiving renal replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Hemofilter lifetime | at day 1

SECONDARY OUTCOMES:
Hemofilter clotting risk factors | at day 1
hemofiltration duration | at day 1
down time value | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France